CLINICAL TRIAL: NCT00004162
Title: Phase I Trial of Liposomal Doxorubicin (Doxil) Based Combination Chemotherapy Regimen in AIDS-Associated Non-Hodgkin's Lymphoma
Brief Title: Liposomal Doxorubicin Plus Combination Chemotherapy in Treating Patients With AIDS-Associated Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067402; UAB-9708; UAB-F970529007; NCI-G99-1627
Record Dates: First submitted 1999-12-10; First posted 2004-08-05 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Lymphoma
Keywords: AIDS-related diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related small noncleaved cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related lymphoblastic lymphoma
MeSH Terms: conditions — Lymphoma | interventions — sargramostim; Methotrexate; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Dose group 1 - dose 1 of Doxorubicin HCL Liposome (Experimental): Patients receive doxorubicin HCl liposome IV, vincristine IV, and methotrexate intrathecally on day 1, followed by oral prednisone on days 1-5. Sargramostim (GM-CSF) is administered subcutaneously on days 5-14 until blood counts recover. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of doxorubicin HCl liposome until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicity. Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter
  Interventions: Biological: sargramostim; Drug: methotrexate; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: vincristine sulfate
- Dose group 2 - dose 2 of Doxorubicin HCL Liposome (Experimental): Patients are stratified by risk group (good vs poor). Patients receive doxorubicin HCl liposome IV, vincristine IV, and methotrexate intrathecally on day 1, followed by oral prednisone on days 1-5. Sargramostim (GM-CSF) is administered subcutaneously on days 5-14 until blood counts recover. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of doxorubicin HCl liposome until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicity. Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter
  Interventions: Biological: sargramostim; Drug: methotrexate; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: vincristine sulfate
- Dose Group 3 - dose 3 of Doxorubicin HCL Liposome (Experimental): Patients are stratified by risk group (good vs poor). Patients receive doxorubicin HCl liposome IV, vincristine IV, and methotrexate intrathecally on day 1, followed by oral prednisone on days 1-5. Sargramostim (GM-CSF) is administered subcutaneously on days 5-14 until blood counts recover. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of doxorubicin HCl liposome until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicity. Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter
  Interventions: Biological: sargramostim; Drug: methotrexate; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: vincristine sulfate
- Dose group 4 - dose 4 of Doxorubicin HCL Liposome (Experimental): Patients are stratified by risk group (good vs poor). Patients receive doxorubicin HCl liposome IV, vincristine IV, and methotrexate intrathecally on day 1, followed by oral prednisone on days 1-5. Sargramostim (GM-CSF) is administered subcutaneously on days 5-14 until blood counts recover. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of doxorubicin HCl liposome until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicity. Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter
  Interventions: Biological: sargramostim; Drug: methotrexate; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: vincristine sulfate
- Dose group 5 - dose 5 of Doxorubicin HCL Liposome (Experimental): Patients are stratified by risk group (good vs poor). Patients receive doxorubicin HCl liposome IV, vincristine IV, and methotrexate intrathecally on day 1, followed by oral prednisone on days 1-5. Sargramostim (GM-CSF) is administered subcutaneously on days 5-14 until blood counts recover. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of doxorubicin HCl liposome until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicity. Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter
  Interventions: Biological: sargramostim; Drug: methotrexate; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: vincristine sulfate
- Dose group 6 - dose 6 of Doxorubicin HCL Liposome (Experimental): Patients are stratified by risk group (good vs poor). Patients receive doxorubicin HCl liposome IV, vincristine IV, and methotrexate intrathecally on day 1, followed by oral prednisone on days 1-5. Sargramostim (GM-CSF) is administered subcutaneously on days 5-14 until blood counts recover. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of doxorubicin HCl liposome until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicity. Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter
  Interventions: Biological: sargramostim; Drug: methotrexate; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: vincristine sulfate
- Dose group 7 - dose 7 of Doxorubicin HCL Liposome (Experimental): Patients are stratified by risk group (good vs poor). Patients receive doxorubicin HCl liposome IV, vincristine IV, and methotrexate intrathecally on day 1, followed by oral prednisone on days 1-5. Sargramostim (GM-CSF) is administered subcutaneously on days 5-14 until blood counts recover. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of doxorubicin HCl liposome until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicity. Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter
  Interventions: Biological: sargramostim; Drug: methotrexate; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: vincristine sulfate
- MTD group (Experimental): Patients are stratified by risk group (good vs poor). Patients receive doxorubicin HCl liposome IV, vincristine IV, and methotrexate intrathecally on day 1, followed by oral prednisone on days 1-5. Sargramostim (GM-CSF) is administered subcutaneously on days 5-14 until blood counts recover. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of doxorubicin HCl liposome until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicity. Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter
  Interventions: Biological: sargramostim; Drug: methotrexate; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: vincristine sulfate

INTERVENTIONS:
Biological: sargramostim
Drug: methotrexate
Drug: pegylated liposomal doxorubicin hydrochloride
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of liposomal doxorubicin plus combination chemotherapy in treating patients who have AIDS-associated non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity and maximum tolerated dose of doxorubicin HCl liposome when administered with combination chemotherapy in patients with AIDS-associated non-Hodgkin's lymphoma. II. Determine the optimal phase II dose of doxorubicin HCl liposome to be administered with the combination chemotherapy regimen. III. Determine the effect of this regimen on HIV viral load in these patients. IV. Determine the clinical response to this regimen by these patients.

OUTLINE: This is a dose escalation study of doxorubicin HCl liposome. Patients are stratified by risk group (good vs poor). Patients receive doxorubicin HCl liposome IV, vincristine IV, and methotrexate intrathecally on day 1, followed by oral prednisone on days 1-5. Sargramostim (GM-CSF) is administered subcutaneously on days 5-14 until blood counts recover. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of doxorubicin HCl liposome until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicity. Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A minimum of 42-48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven good or poor prognosis AIDS-associated non-Hodgkin's lymphoma expressing CD20 antigen HIV positive Stage II-IV Good risk patients are defined as: Karnofsky 80-100% No prior history of AIDS defining illness No bone marrow involvement with lymphoma No clinical, radiographic, or cytologic evidence of CNS lymphoma Bidimensionally measurable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 80-100% Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count greater than 1,000/mm3 Platelet count greater than 75,000/mm3 Hemoglobin greater than 9 g/dL Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT or SGPT less than 5 times ULN Alkaline phosphatase less than 5 times ULN Renal: Creatinine no greater than 1.5 times ULN Other: Not pregnant No active opportunistic or any other serious infection No other malignancy (including any other AIDS-associated malignancy) except stable cutaneous Kaposi's sarcoma No serious medical or psychiatric condition

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior doxorubicin or doxorubicin HCl liposome No prior chemotherapy for non-Hodgkin's lymphoma, except single dose of intrathecal chemotherapy at time of staging lumbar puncture Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: At least 2 weeks since major surgery Other: No concurrent treatment for Kaposi's sarcoma Concurrent antiretroviral therapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 1997-06; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
Determine the toxicity and maximum tolerated dose of doxorubicin HCl liposome when administered with combination chemotherapy in patients with AIDS-associated non-Hodgkin's lymphoma. | baseline to last dose of study drug

SECONDARY OUTCOMES:
Determine the optimal phase II dose of doxorubicin HCl liposome to be administered with the combination chemotherapy regimen. | baseline to last dose of study drug
Determine the effect of this regimen on HIV viral load in these patients | baseline to survival
Determine the clinical response to this regimen by these patients | baseline to survival

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor N. Saleh, MD, Study Chair — University of Alabama at Birmingham
Locations (1):
- University of Alabama Comprehensive Cancer Center, Birmingham, Alabama, United States